CLINICAL TRIAL: NCT02399722
Title: Prospective Randomized Trial Comparing the Combination of a Polymeric Membrane Dressing Plus Negative Pressure Wound Therapy Against Negative Pressure Wound Therapy Alone: The WICVAC Study
Brief Title: Combination of a Polymeric Membrane Dressing Plus Negative Pressure Wound Therapy Against Negative Pressure Wound Therapy Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilhelminenspital Vienna (Other)
Responsible Party: Principal Investigator, Edda Skrinjar, M.D., M.D., Wilhelminenspital Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WICVAC 1.0
Record Dates: First submitted 2015-03-22; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Wound
Keywords: Negative Pressure Wound Therapy, polymeric membrane dressing, wounds
MeSH Terms: conditions — Wounds and Injuries | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAC mono therapy (Active Comparator): negative pressure wound therapy alone
  Interventions: Device: VAC mono therapy
- WICVAC combined therapy (Active Comparator): Polymeric membrane dressing combined with negative pressure wound therapy
  Interventions: Device: WICVAC

INTERVENTIONS:
Device: WICVAC — combined wound therapy
  Other Names: Polymeric membrane dressing (PolyMem® WIC)
  Arms: WICVAC combined therapy
Device: VAC mono therapy — mono therapy
  Other Names: NPWT (VAC)
  Arms: VAC mono therapy

SUMMARY:
In surgical units negative pressure wound therapy (NPWT) is often used to facilitate wound healing. The recommended frequency of change every third to fourth day causes an immense workload.

The purpose of this study is to evaluate the effect of an additional polymeric membrane interface dressing (PolyMem® WIC) as primary wound contact layer in NPWT in comparison to NPWT alone on the number of required dressing changes until wound closure as the primary endpoint. Secondary endpoints are: time to heal and wound associated pain.

DETAILED DESCRIPTION:
Background:

The treatment of chronic wounds requires time and resources. Optimized resource utilization in treatment of chronic wounds is of medical and economic interest.

Negative pressure wound therapy (NPWT) is widely used for the treatment of chronic wounds and surgical site infections. NPWT is indicated for the treatment of diabetic leg ulcers, lower leg ulcers as a result of peripheral arterial occlusive disease, pressure wounds, surgical incisional wounds, traumatic wounds, burns, infected wounds, necrotizing fasciitis, infected sternal wounds, and after skin grafting to facilitate healing. The polyurethane foam of the NPWT is directly applied to a wound bed and sealed with a transparent occlusive film prior to application of a negative pressure at 75 to 125 mmHg continuous suction. Prolonged placement of the foam in the wound bed results in tissue ingrowth. Then, removal of the foam becomes increasingly difficult and is often accompanied by pain, bleeding, and traumatization of the healing wound. Therefore, various efforts have been made to decrease wound tissue damage and pain during dressing change, including the use of different primary wound fillers, administration of topical analgesics or placement of various interface dressings. Yet, the effect of a non-adherent polymeric interface dressing on wearing time and frequency of dressing changes has not been studied.

Methods:

Sixty consecutive patients with chronic wounds of lower extremities or surgical site infections after revascularization are randomly allocated to either treatment with conventional negative pressure wound therapy (VAC arm, control) or negative pressure wound therapy with additional polymeric interface dressing (VAC + PolyMem® WIC, WICVAC, study arm). The polymeric membrane dressing is applied as direct wound contact layer, covered with the polyurethane foam dressing of the NPWT. The pink polymeric membrane dressing, which is left partially visible at the margin of the wound bed under the black polyurethane foam, serves as color indicator for the time-point of dressing change upon loss of the pink color. Patient characteristics, wound size at each dressing change, pain during treatment and the number of dressing changes needed until wound closure are documented.

Statistical analysis Sample size estimation was based on detecting a 20% difference in the number of dressing changes in favor of the WICVAC - study arm, with a type I error of 0.05 and type II error of 0.2. At least 23 patients are required for each study arm. Data are analyzed for statistical distribution. Due to skewed data distribution Mann-Whitney-U tests are applied for assessment of differences in primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* presence of a chronic wound or an infected wound with adequate perfusion
* successful revascularization of underlying PAOD or diabetic macroangiopathy of lower extremities within 24-48 h before study allocation

Exclusion Criteria:

* unfeasible or unsuccessful revascularization
* preexisting documented allergies against used products
* refusal of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of dressing changes | 30 days
  number of dressing changes until wound closure

SECONDARY OUTCOMES:
Pain | 30 days
  pain during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Assadian, PD MD, Principal Investigator — Department of Vascular and Endovascular Surgery - Wilhelminenhospital